CLINICAL TRIAL: NCT01189968
Title: A Phase 1b Study of Carboplatin and Pemetrexed Plus Demcizumab (OMP-21M18) as 1st-line Treatment in Subjects With Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Carboplatin and Pemetrexed Plus Demcizumab (OMP-21M18) in Subjects With Non-Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M18-004
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Phase 1,; dose escalation,; histologically; confirmed; malignancy; metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Neoplasm Metastasis | interventions — demcizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carboplatin and Pemetrexed plus demcizumab (Experimental): Carboplatin and Pemetrexed plus demcizumab
  Interventions: Drug: Demcizumab
- Pemetrexed plus demcizumab (Experimental): Pemetrexed plus demcizumab
  Interventions: Drug: Demcizumab

INTERVENTIONS:
Drug: Demcizumab — The 6 subjects in the first cohort will receive demcizumab 5 mg/kg once every 3 weeks; the 6 subjects in the subsequent cohort will be treated with 10 mg/kg once every 3 weeks; and the 6 subjects in the final cohort will be treated with 15 mg/kg once every 3 weeks. A Data Safety Monitoring Board (DSMB) will review the data for the 6 subjects in each dose cohort after the last subject in that cohort has been on study for 56 days and then decide whether it is safe to escalate to the next highest dose cohort. Once the dose-escalation portion of the study has been completed, 14 additional subjects will be treated at the highest dose level that the DSMB deems as safe.
  Other Names: OMP-21M18

SUMMARY:
The purpose of this study is to test the safety and determine the optimal dose of a new drug, demcizumab (OMP-21M18), when given in combination with carboplatin and pemetrexed, a standard drug treatment regimen for non-squamous non-small cell lung cancer (NSCLC). Participants must not have received prior chemotherapy for their NSCLC. Demcizumab is a humanized monoclonal antibody (a protein made in the laboratory) developed to target cancer stem cells. The way the body handles demcizumab will also be investigated.

Up to 50 subjects will be enrolled at up to 8 centers in Australia, New Zealand, and Spain. Up to 28 days (4 weeks) prior to treatment you will undergo testing to determine your eligibility to take part in this study, and then if enrolled in the study you will receive intravenous (in the vein) infusions of the demcizumab, carboplatin, and pemetrexed administered on the same day, every 21 days for 4 cycles, or until it has been shown that your cancer has progressed. If your physician decides to delay treatment with one of the agents due to side effects, the other agents may still be administered as scheduled. After 4 cycles, if you have stable or improved disease, you will continue to receive pemetrexed once every 21 days as maintenance therapy. You will undergo assessments every 8 weeks to determine the status of your disease.

DETAILED DESCRIPTION:
Current cancer therapies often produce an initial reduction in tumour size but may not have longterm benefits. One possible explanation for this is the presence of cancer cells known as cancer stem cells. Cancer stem cells represent a small part of the tumour but are believed to be responsible for much of the growth and spread of the cancer. They may also be more resistant to traditional therapy, such as chemotherapy and radiation therapy.

Up to 50 subjects will be enrolled at up to 8 centers in Australia, New Zealand, and Spain. Up to 28 days (4 weeks) prior to treatment you will undergo testing to determine your eligibility to take part in this study, and then if enrolled in the study you will receive intravenous (in the vein) infusions of the demcizumab, carboplatin, and pemetrexed administered on the same day, every 21 days for 4 cycles, or until it has been shown that your cancer has progressed. If your physician decides to delay treatment with one of the agents due to side effects, the other agents may still be administered as scheduled. After 4 cycles, if you have stable or improved disease, you will continue to receive pemetrexed once every 21 days as maintenance therapy. You will undergo assessments every 8 weeks to determine the status of your disease.

In addition to routine testing of blood and urine (for complete blood counts with differential and platelets, coagulation studies to determine how quickly your blood is clotting; serum chemistries; B-type natriuretic peptide [BNP] and Troponin I, which indicate how well your heart if working; creatinine clearance to measure your kidney function and urinalysis), special tests will be performed during the study at specific time points.

In addition, you will have an ECG and doppler echocardiogram performed during screening, then every 28 days on study and at treatment termination. Your Doppler echocardiograms may be sent to a Cardiologist at another hospital who may perform a central read on some of the doppler echocardiograms in this study. Finally, you will have a head CT or MRI at baseline and CT scans and/or other radiographs performed every 56 days to assess the status of your tumor.

The study includes an optional part which will investigate how variations in people's genetic makeup affect their response to medications. This involves the collection of one blood sample just before participants receive their first dose of study treatment. DNA will be extracted from the blood sample for testing.

ELIGIBILITY:
Inclusion criteria

1. Subjects must have histologically confirmed unresectable, locally advanced, recurrent, or metastatic non-squamous NSCLC. Subjects may not have received prior therapy for their unresectable, locally advanced, recurrent, or metastatic non-squamous NSCLC. Subjects may have received prior surgery, prior radiotherapy, and/or prior neoadjuvant or adjuvant chemotherapy (they must have discontinued prior neoadjuvant or adjuvant chemotherapy at least 12 weeks prior to study entry).
2. Age >21 years
3. ECOG performance status <2 (see Appendix B)
4. Life expectancy of more than 3 months
5. Subjects must have normal organ and marrow function as defined below:

   * Leukocytes >3.5 x 109/L
   * Absolute neutrophil count >1.25 x 109/L Hemoglobin >100 g/L
   * Platelets >125 X 109/L
   * Total bilirubin <2 X institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) <5 X institutional ULN
   * Alkaline phosphatase <5 X institutional ULN
   * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) within institutional ULN
   * Calculated creatinine clearance >60 mL/min using the Cockcroft and Gault formula as follows:

   Creatinine clearance (mL/min) = (140 - age) x ideal body weight [kg] 0.814 x serum creatinine [μmol/L] For women multiply the value from the equation above by 0.85. Where age is in years, weight is in kg, and serum creatinine is in μmol/L.
6. Women of childbearing potential must have had a prior hysterectomy or have a negative serum pregnancy test and be using adequate contraception prior to study entry and must agree to use adequate contraception from study entry through at least 6 months after discontinuation of study drugs. Men must also agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and from study entry through at least 6 months after discontinuation of study drugs. Should a woman enrolled in the study or a female partner of a man enrolled in the study become pregnant or suspect she is pregnant while participating in this study or within 6 months after discontinuation of the study drugs, the Investigator should be informed immediately.
7. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria

Subjects who meet any of the following criteria will not be eligible for participation in the study:

1. Subjects receiving any other investigational agents or anti-cancer therapy.
2. Subjects with brain metastases (subjects must have a CT scan or MRI of the head within 28 days prior to enrollment to rule out brain metastases), uncontrolled seizure disorder, or active neurologic disease
3. History of a significant allergic reaction attributed to humanized or human monoclonal antibody therapy
4. Significant intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
5. Pregnant women or nursing women
6. Subjects with known HIV infection
7. Known bleeding disorder or coagulopathy
8. Subjects receiving heparin, warfarin, or other similar anticoagulants. Note: Subjects may be receiving low-dose aspirin and/or non-steroidal anti-inflammatory agents.
9. Subjects with known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease
10. New York Heart Association Classification II, III, or IV (See Appendix D)
11. Subjects with a blood pressure of >140/90 mmHg. The BP should be taken using the method described in Section 9.3. Subjects taking antihypertensive medications must be taking ≤ 2 medications to obtain this level of BP control.
12. Subjects with metastases that are currently involving the lumen of the gastrointestinal tract
13. Subjects with squamous cell carcinoma of the lung
14. Subjects with recent (within the last 8 weeks) hemoptysis >2.5 mL and subjects with serious bleeding from another site within this timeframe
15. Subjects with current evidence of cardiac ischemia or heart failure within the last 6 months, subjects who are receiving any medications for cardiac ischemia, subjects with a B-type natriuretic peptide (BNP) value of >100 pg/mL, subjects with a LVEF <50%, subjects with pulmonary hypertension defined as a peak tricuspid velocity >3.4 m/s on doppler echocardiogram or subjects that have received a total cumulative dose of ≥400 mg/m2 doxorubicin.
16. Subjects with ECG evidence of ischemia or ≥ Grade 2 ventricular arrhythmia, subjects who have a history of acute myocardial infarction within 6 months, or subjects with unstable angina.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To the determine the maximum tolerated dose of demcizumab (OMP-21M18) plus carboplatin and pemetrexed | When each patient in the dose cohort reaches Day 56

SECONDARY OUTCOMES:
To determine the safety of carboplatin and pemetrexed plus demcizumab (OMP-21M18) | until treatment termination plus 30 days
To determine the rates of immunogenicity of carboplatin and pemetrexed plus demcizumab (OMP-21M18) | Up to 12 weeks post treatment termination
To determine the preliminary efficacy of carboplatin and pemetrexed plus demcizumab (OMP-21M18) | Until disease progression
To determine population pharmacokinetics | Day 21 and 63
To determine the exploratory biomarker changes of carboplatin and pemetrexed plus demcizumab (OMP-21M18) | Until Day 112

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (4):
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- New Zealand (2):
  - Auckland Hospital, Grafton, Auckland
  - Waikato Hospital, Hamilton
- START Madrid, Madrid, Spain

REFERENCES:
- [Derived] McKeage MJ, Kotasek D, Markman B, Hidalgo M, Millward MJ, Jameson MB, Harris DL, Stagg RJ, Kapoun AM, Xu L, Hughes BGM. Phase IB Trial of the Anti-Cancer Stem Cell DLL4-Binding Agent Demcizumab with Pemetrexed and Carboplatin as First-Line Treatment of Metastatic Non-Squamous NSCLC. Target Oncol. 2018 Feb;13(1):89-98. doi: 10.1007/s11523-017-0543-0. PMID 29188408